CLINICAL TRIAL: NCT04980027
Title: Multicentre Phase IV Single Arm Clinical Trial to evaluAte the saFety and Efficacy of Gla-300 in insUlin-naïve Patients With Type 2 DiAbetes uncontRolled on Oral Antihyperglycemic Drugs
Brief Title: Evaluation of the Safety and Efficacy of Insulin Glargine 300 U/ml (Gla-300) in Insulin-naïve Patients With Type 2 Diabetes Mellitus Uncontrolled on Oral Antihyperglycemic Drugs
Acronym: SAFEGUARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS16665; U1111-1255-5143 (Other: UTN)
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insuline Glargine (U300) (Gla-300) (Experimental): Insulin glargine (U300) once daily for 24 weeks on top of non-insulin antidiabetic drug. Insulin dose will be adjusted according to the recommended titration algorithm
  Interventions: Drug: Insulin glargine (U300)

INTERVENTIONS:
Drug: Insulin glargine (U300) — Pharmaceutical form:Solution for injection in a prefilled pen Route of administration: Subcutaneous
  Other Names: HOE901 Toujeo

SUMMARY:
Primary Objective:

To evaluate the safety of Gla-300 in insulin naïve T2D participants uncontrolled on oral antihyperglycemic drugs

Secondary Objective:

To assess the efficacy of Gla-300 on glycemic control in insulin naïve T2D participants uncontrolled on oral anti-hyperglycemic drugs To assess change in participant's treatment satisfaction using DTSQs (Diabetes Treatment Satisfaction Questionnaire)

DETAILED DESCRIPTION:
The maximum study duration per participant is 27 weeks including a screening period of up to 2 weeks, a 24-week treatment period and a post-treatment follow-up phone call visit after 3 days after the end of treatment.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 diabetes mellitus
* Participants who are insulin naïve on at least one oral antihyperglycemic drug (metformin,sulfonylurea, thiazolidinedione, DPP-4 inhibitor, SGLT-2 inhibitor, glinide, α-glucosidase inhibitor) with or without glucagon-like peptide 1 receptor agonists (GLP-1 RAs) for a minimum period of 6 months prior to screening.
* HbA1c between 7.5% (58 mmol/mol) and 10% (86 mmol/mol) inclusive, during screening.

Exclusion criteria:

* History of severe hypoglycemia requiring emergency room admission or hospitalization within 3 months prior to screening visit.
* Proliferative retinopathy or maculopathy requiring treatment according to the Investigator
* Treatment with any insulin including basal insulin, mixed insulin (premixes), rapid insulin, and fast-acting insulin analogues in the last 6 months before screening visit (use ≤10 days in relation to hospitalization or an acute illness is accepted).
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for 2 weeks or more within 8 weeks prior to screening visit.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Treatment Emergent Adverse Events (TEAEs) | Baseline to Week 24
  TEAEs including serious adverse events (SAEs) and hypoglycemic episode

SECONDARY OUTCOMES:
Percentage of participants with at least one confirmed hypoglycemia event | Baseline to Week 24
Change in HbA1c from Baseline to week 12 and week 24 | Baseline to Week 12 and Week 24
Percentage of participants reaching HbA1c target of <7% | Week 12 and Week 24
Percentage of participants reaching targeted fasting self-monitored blood glucose (SMBG) of 80 to 110 mg/dL (4.4 to 6.1 mmol/L) | Week 12 and Week 24
Change in fasting plasma glucose (FPG) from Baseline to Week 24 | Baseline to Week 24
Change in fasting SMBG from Baseline to Week 24 | Baseline to Week 24
Change in 7-point SMBG profile from Baseline to Week 24 | Baseline to Week 24
Percentage of participants requiring rescue therapy | Week 12 and Week 24
Change in body weight from Baseline to Week 12 and Week 24 | Baseline to Week 12 and Week 24
Change in insulin dose from Baseline to Week 12 and Week 24 | Baseline to Week 12 and Week 24
Change in DTSQs scores from Baseline to Week 12 and Week 24 | Baseline to Week 12 and Week 24
  The Diabetes Treatment Satisfaction Questionnaire - status version (DTSQs) is measuring patients' satisfaction with their diabetes treatment.Total treatment satisfaction score range from 0 (no satisfaction) to 36 (improvement in treatment satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- India (2):
  - Investigational site Number 3560003, Jaipur
  - Investigational site Number 3560013, Nashik

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Mohan V, Sethi B, Jain SM, Sahay R, Ramanathan B, Murthy S, Singh KP, Menon S, Gadekar A, Salvi V, Gandhi K. Multicenter, Phase 4 Clinical Study from India to Evaluate the Safety and Efficacy of Insulin Glargine 300 U/ml in Insulin-Naive People with Type 2 Diabetes Uncontrolled on Oral Anti-hyperglycemic Drugs: SAFEGUARD Study. Diabetes Ther. 2025 Jul;16(7):1367-1383. doi: 10.1007/s13300-025-01736-5. Epub 2025 May 8. PMID 40338497
- See also: LPS16665 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25286&tenant=MT_SNY_9011